CLINICAL TRIAL: NCT00682019
Title: A Randomized, Double-Blind, Parallel-Group, Placebo-Controlled Study Evaluating the Duration of Efficacy and Safety of Vardenafil Administered for 10 Weeks in a Flexible-Dose Regimen Compared to Placebo in Subjects With Erectile Dysfunction
Brief Title: Study Evaluation the Efficacy and Safety of Vardenafil in Subjects With Erectile Dysfunction for 10 Weeks
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 100493
Record Dates: First submitted 2008-04-18; First posted 2008-05-21 (Estimated); Last update posted 2013-10-14 (Estimated); Status verified 2013-10

CONDITIONS: Erectile Dysfunction
Keywords: Erectile Dysfunction; Vardenafil
MeSH Terms: conditions — Erectile Dysfunction | interventions — Vardenafil Dihydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Levitra (Vardenafil, BAY38-9456)
- Arm 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levitra (Vardenafil, BAY38-9456) — 5mg, 10mg or 20mg taken 8 hours before sexual intercourse
  Arms: Arm 1
Drug: Placebo — matching placebo
  Arms: Arm 2

SUMMARY:
The aim of this international study was to determine if 10 weeks of flexible-dose vardenafil therapy demonstrates superior efficacy compared to the dummy drug (placebo) in Erectile dysfunction subjects of a broad etiology when dosed 8 (+/-2) hours prior to sexual intercourse. In addition it should have been determined, if subjects with ED from a broad etiology can tolerate 10 weeks of flexible-dose vardenafil therapy when dosed 8(+/-2) hours prior to sexual intercourse.

ELIGIBILITY:
Inclusion Criteria:

* Men >/= 18 years of age, with 6 months or longer diagnosis of ED as defined by NIH Consensus statement,
* History of unresponsiveness to sildenafil
* Stable sexual relationship for > 6 month.

Exclusion Criteria:

* Primary hypoactive sexual desire
* History of myocardial infarction, stroke or life-threatening arrhythmia within prior 6 month
* Nitrate therapy.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 383 (Actual)
Dates: Start 2003-12; Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
Per-patient success rates based on Sexual Encounter Profile, Question 3 | 10 weeks

SECONDARY OUTCOMES:
Per-subject success rates based on Sexual Encounter Profile, Question 2 | 10 weeks
International Index of Erectile Function- Erectile Function domain score | 10 weeks
Global Assessment Question (GAQ) | 10 weeks
Safety and tolerability | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer